CLINICAL TRIAL: NCT01920061
Title: A PHASE 1B OPEN-LABEL THREE-ARM MULTI-CENTER STUDY TO ASSESS THE SAFETY AND TOLERABILITY OF PF-05212384 (PI3K/MTOR INHIBITOR) IN COMBINATION WITH OTHER ANTI-TUMOR AGENTS
Brief Title: A Study Of PF-05212384 In Combination With Other Anti-Tumor Agents and in Combination With Cisplatin in Patients With Triple Negative Breast Cancer in an Expansion Arm (TNBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B2151002; 2013-001390-24 (EudraCT Number)
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Neoplasm
Keywords: Advanced cancer; solid tumors; PI3K; mTOR; PI3K/mTOR; metastatic; Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms | interventions — gedatolisib; Docetaxel; Cisplatin; dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A (Experimental)
  Interventions: Drug: PF-05212384 (gedatolisib); Drug: Docetaxel
- Arm B (Experimental)
  Interventions: Drug: PF-05212384 (gedatolisib); Drug: Cisplatin
- Arm C (Experimental)
  Interventions: Drug: PF-05212384 (gedatolisib); Drug: Dacomitinib
- Expansion Arm 1 (Experimental)
  Interventions: Drug: PF-05212384 (gedatolisib); Drug: Cisplatin
- Expansion Arm 2 (Experimental)
  Interventions: Drug: PF-05212384 (gedatolisib); Drug: Cisplatin

INTERVENTIONS:
Drug: PF-05212384 (gedatolisib) — PF-05212384 weekly intravenous infusions starting at 90 mg/wk as a 3 week cycle
Drug: Docetaxel — Docetaxel intravenous infusions once every 3 weeks starting at 75 mg/m^2
  Arms: Arm A
Drug: Cisplatin — Cisplatin intravenous infusions once every 3 weeks starting at 75 mg/m^2
  Arms: Arm B; Expansion Arm 1; Expansion Arm 2
Drug: Dacomitinib — Dacomitinib to be taken orally as a continuous once daily regimen at a starting dose of 30 mg
  Arms: Arm C

SUMMARY:
This study will evaluate PF-05212384 (gedatolisib) PI3K/mTOR inhibitor)) in combination with either docetaxel, cisplatin or dacomitinib in select advanced solid tumors. The study will assess the safety, pharmacokinetics and pharmacodynamics of these combinations in patients with advanced cancer in order to determine the maximum tolerated dose in each combination. The cisplatin combination expansion portion will evaluate the anti tumor activity of PF 05212384 plus cisplatin in patients with TNBC in 2 separate Arms (Arm 1 and Arm 2).

ELIGIBILITY:
Inclusion Criteria:

Cisplatin Combination Expansion:

Arm 1:Patients with TNBC with no prior cytotoxic chemotherapy therapy in the metastatic setting; Arm 2: Patients with TNBC and one or two prior cytotoxic therapies in the metastatic setting.

* Arm A: castrate resistant prostate cancer, advanced breast cancer, or non-small cell lunch cancer that are candidates for treatment with a docetaxel-based combination.
* Arm B: Urothelial transitional cell cancer, triple negative breast cancer, ovarian cancer or non small cell lunch cancer that are candidates for a cisplatin-based combination.
* Arm C: Her2+ breast cancer refractory to prior herceptin or lapatinib, her2+ esophagal-gastric cancer, head and neck squamous cell cancer, or non small cell lunch cancer that are candidates for treatment with a dacomitinib-based combination.
* Availability of archival tumor biopsy sample or willing to provide fresh biopsy if not available.
* Eastern Cooperative Oncology Group [ECOG] performance must be 0 or 1.
* Adequate bone marrow, renal and liver function.

Exclusion Criteria:

* Prior therapy for Cisplatin Combination Expansion:

  * Prior platinum (carboplatin or cisplatin) in either the adjuvant or metastatic setting;
  * Prior radiation to >25% bone marrow as estimated by the Investigator.
* Patients with known symptomatic brain metastases.
* Chemotherapy, radiotherapy, biologics or investigational agent within 4 weeks of the lead-in dose.
* Major surgery within 4 weeks of the baseline disease assessments.
* >2 prior regimens containing cytotoxic chemotherapy in the metastatic setting.
* Active bacterial, fungal or viral infection.
* Uncontrolled or significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - Westwood Bowyer Clinic, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Santa Monica UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA Hematology Oncology, Santa Monica, California
  - University of Colorado Denver CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Harper Professional Building, Detroit, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina/ University Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC SCTR Research, Charleston, South Carolina
  - MUSC Health East Cooper, Mt. Pleasant, South Carolina
  - MUSC Specialty Care-North, North Charleston, South Carolina
- Canada (2):
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
- Italy (2):
  - Istituto Europeo di Oncologia - Divisione Sviluppo di Nuovi Farmaci per Terapie Innovative, Milan, MI
  - Istituto Regina Elena Struttura Complessa Oncologia Medica A, Roma, RM
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - University College London Hospital, NIHR UCLH Clinical Research Facility, London
  - Oxford Cancer Centre, Oxford

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Curigliano G, Shapiro GI, Kristeleit RS, Abdul Razak AR, Leong S, Alsina M, Giordano A, Gelmon KA, Stringer-Reasor E, Vaishampayan UN, Middleton M, Olszanski AJ, Rugo HS, Kern KA, Pathan N, Perea R, Pierce KJ, Mutka SC, Wainberg ZA. A Phase 1B open-label study of gedatolisib (PF-05212384) in combination with other anti-tumour agents for patients with advanced solid tumours and triple-negative breast cancer. Br J Cancer. 2023 Jan;128(1):30-41. doi: 10.1038/s41416-022-02025-9. Epub 2022 Nov 5. PMID 36335217
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2151002&StudyName=A%20Study%20Of%20PF-05212384%20In%20Combination%20With%20Other%20Anti-Tumor%20Agents

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Arm A included 5 sub-arms: Arms A1, A2, A3, A4, A5 Arm B included 8 sub-arms: Arms B1, B2, B3, B4, B5, B6, B7, B8 Arm C included 5 sub-arms: Arms C1, C1h, C2, C3, C4 Arm B Expansion included 2 sub-arms: Arms 1, 2
Pre-assignment Details: A total of 110 subjets were enrolled in this study and 3 of them didn't received any study treatment.
Groups:
- Arm A1: 90 mg PF-05212384 + Docetaxel: Participants with castrate resistant prostate cancer (CRPC), advanced breast cancer (ABC), or non-small cell lung cancer (NSCLC) that were candidates to treatment with a docetaxel-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90 mg once on Day -7 and Cycle 1 Day 2, and docetaxel 75 mg/m2 1-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received docetaxel 75 mg/m2 1-hour IV infusion once followed by PF-05212384 90 mg once. The maximum duration of PF-05212384 treatment was 505 days and the maximum duration of docetaxel treatment was 445 days.
- Arm A2: 110 mg PF-05212384 + Docetaxel: Participants with CRPC, ABC, or NSCLC that were candidates to treatment with a docetaxel-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 110 mg once on Day -7 and Cycle 1 Day 2, and docetaxel 75 mg/m2 1-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received docetaxel 75 mg/m2 1-hour IV infusion once followed by PF-05212384 110 mg once. The maximum duration of PF-05212384 treatment was 505 days and the maximum duration of docetaxel treatment was 445 days.
- Arm A3: 130 mg PF-05212384 + Docetaxel: Participants with CRPC, ABC, or NSCLC that were candidates to treatment with a docetaxel-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 130 mg once on Day -7 and Cycle 1 Day 2, and docetaxel 75 mg/m2 1-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received docetaxel 75 mg/m2 1-hour IV infusion once followed by PF-05212384 130 mg once. The maximum duration of PF-05212384 treatment was 505 days and the maximum duration of docetaxel treatment was 445 days.
- Arm A4: 150 mg PF-05212384 + Docetaxel: Participants with CRPC, ABC, or NSCLC that were candidates to treatment with a docetaxel-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 150 mg once on Day -7 and Cycle 1 Day 2, and docetaxel 75 mg/m2 1-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received docetaxel 75 mg/m2 1-hour IV infusion once followed by PF-05212384 150 mg once. The maximum duration of PF-05212384 treatment was 505 days and the maximum duration of docetaxel treatment was 445 days.
- Arm A5: 180 mg PF-05212384 + Docetaxel: Participants with CRPC, ABC, or NSCLC that were candidates to treatment with a docetaxel-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 180 mg once on Day -7 and Cycle 1 Day 2, and docetaxel 75 mg/m2 1-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received docetaxel 75 mg/m2 1-hour IV infusion once followed by PF-05212384 180 mg once. The maximum duration of PF-05212384 treatment was 505 days and the maximum duration of docetaxel treatment was 445 days.
- Arm B1: 90 mg PF-05212384 + Cisplatin: Participants with urothelial transitional cell cancer (TCC), triple negative breast cancer (TNBC), NSCLC or ovarian cancer (OC) that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 90 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B2: 110 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 110 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 110 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B3: 130 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 130 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 130 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B4: 150 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 150 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 150 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B5: 180 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 180 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 180 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B6: 215 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 215 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 215 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B7: 260 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 260 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 260 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm B8: 310 mg PF-05212384 + Cisplatin: Participants with TCC, TNBC, NSCLC or OC that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 310 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 310 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm C1: 90 mg PF-052123 84 + 30 mg Dacomitinib: Participants with Her2+ breast cancer (BC) refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, head and neck squamous cell cancer (HNSCC), or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90 mg once on Day -14 and dacomitinib 30 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 30 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 30 mg orally once followed by PF-05212384 90 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 30 mg orally once followed by PF-05212384 90 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
- Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib: Participants with BC refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, HNSCC, or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90 mg once on Day -14 and dacomitinib 45 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 45 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 45 mg orally once followed by PF-05212384 90 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 45 mg orally once followed by PF-05212384 90 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
- Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib: Participants with BC refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, HNSCC, or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 110 mg once on Day -14 and dacomitinib 30 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 30 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 30 mg orally once followed by PF-05212384 110 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 30 mg orally once followed by PF-05212384 110 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
- Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib: Participants with BC refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, HNSCC, or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 130 mg once on Day -14 and dacomitinib 30 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 30 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 30 mg orally once followed by PF-05212384 130 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 30 mg orally once followed by PF-05212384 130 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
- Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib: Participants with BC refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, HNSCC, or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 150 mg once on Day -14 and dacomitinib 30 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 30 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 30 mg orally once followed by PF-05212384 150 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 30 mg orally once followed by PF-05212384 150 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
- Arm 1: 1L Metastatic: Participants with TNBC with no prior cytotoxic chemotherapy therapy in the metastatic setting received intravenous infusion of cisplatin 75 mg/m2 2-hour IV infusion followed by intravenous infusion of PF-05212384 180 mg. The maximum duration of PF-05212384 treatment was 728 days and the maximum duration of cisplatin treatment was 211 days.
- Arm 2: 2L/3L Metastatic: Participants with TNBC and one or two prior cytotoxic therapies in the metastatic setting received intravenous infusion of cisplatin 75 mg/m2 2-hour IV infusion followed by intravenous infusion of PF-05212384 180 mg. The maximum duration of PF-05212384 treatment was 728 days and the maximum duration of cisplatin treatment was 211 days.
Period: Overall Study
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-052123 84 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastatic | Arm 2: 2L/3L Metastatic
Started | 4 | 5 | 3 | 4 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 3 | 16 | 4 | 7 | 3 | 3 | 10 | 12
Received Treatment | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Completed | 2 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 2 | 1 | 5 | 2 | 1 | 10 | 3 | 4 | 1 | 1 | 4 | 8
Not Completed | 2 | 4 | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 2 | 5 | 3 | 2 | 6 | 1 | 3 | 2 | 2 | 6 | 4
Not completed — Death | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3
Not completed — Other | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 4 | 0 | 1 | 1 | 0 | 1 | 1
Not completed — Participant refused further follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-052123 84 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastatic | Arm 2: 2L/3L Metastatic | Total
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (4.7) | 62.0 (10.9) | 61.7 (7.6) | 58.3 (15.9) | 63.6 (8.1) | 57.3 (9.1) | 51.7 (13.6) | 54.7 (15.9) | 54.0 (9.6) | 55.7 (8.5) | 54.6 (11.1) | 58.2 (13.7) | 59.5 (13.4) | 53.4 (14.1) | 54.3 (22.1) | 55.4 (8.8) | 49.7 (6.4) | 56.3 (12.4) | 52.4 (13.6) | 54.8 (11.6) | 55.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 10 | 3 | 2 | 8 | 4 | 0 | 2 | 1 | 10 | 12 | 73
  Male | 2 | 2 | 2 | 1 | 3 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 7 | 0 | 7 | 1 | 2 | 0 | 0 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 3 | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 9 | 4 | 2 | 14 | 3 | 7 | 2 | 3 | 9 | 11 | 97
  Black | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) - Arms A, B and C
Description: DLT was defined as any of the following adverse events (AEs) attributable to the combination: (1) hematologic: grade 4 neutropenia lasting >7 days; febrile neutropenia; grade >=3 neutropenia with infection; grade 3 thrombocytopenia with bleeding; grade 4 thrombocytopenia; (2) non-hematologic: grade >=2 pneumonitis; grade>=3 toxicities, except pneumonitis, and excluding those that had not been maximally treated; persistent, intolerable toxicities which resulted in the failure to deliver at least 3 of the 4 doses of PF-05212384 for Arms A and B or at least 3 of the 4 doses of PF-05212384 and 75% of dacomitinib for Arm C during the first cycle; the persistent, intolerable toxicities which result in delay of the start of the second cycle by more than 2 weeks relative to the scheduled start; in an asymptomatic participant, the grade 3 QTc prolongation persists after correction of any reversible causes.
Time Frame: Up to 21 days
Population: The per protocol analysis set included all enrolled participants who received at least one dose of study medication and who did not receive less than 75% or more than 125% of the planned Cycle 1 dose of either study drug in the combination.
Measure: Count of Participants; unit: Participants
Groups:
- Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib: Participants with Her2+ breast cancer (BC) refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, head and neck squamous cell cancer (HNSCC), or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90 mg once on Day -14 and dacomitinib 30 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 30 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 30 mg orally once followed by PF-05212384 90 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 30 mg orally once followed by PF-05212384 90 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 2 | 13 | 2 | 7 | 3 | 2
Participants
  With DLT | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0
  No DLT | 4 | 3 | 2 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 8 | 3 | 0 | 13 | 0 | 5 | 3 | 2
  Data missing | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Objective Response - Arm B Expansion
Description: Percentage of participants with objective response based on the assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response.
  Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm) and no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions.
Time Frame: Cycle 1 Day 1 up to 18 months
Population: The response analysis set included all participants who received at least one dose of study medication, had the disease under study, and who had an adequate baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Arm 1: 1L Metastasic: Participants with TNBC with no prior cytotoxic chemotherapy therapy in the metastatic setting received intravenous infusion of cisplatin 75 mg/m2 2-hour IV infusion followed by intravenous infusion of PF-05212384 180 mg. The maximum duration of PF-05212384 treatment was 728 days and the maximum duration of cisplatin treatment was 211 days.
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 12
Percentage of participants | 40.0 [12.2 to 73.8] | 33.3 [9.9 to 65.1]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causality) - Arms A, B, C and B Expansion
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participants administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. Treatment Emergent AEs were those occurred for the first time after the start of study treatment and within 28 days after final dose of study treatment and was not seen prior to the start of treatment, or those were seen prior to the start of study treatment but increased in Common Terminology Criteria for Adverse Events (CTCAE) grade after the start of study treatment and within 28 days after final dose of study treatment. AEs were graded by the investigator according to the CTCAE version 4.03 : Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: From the first dose of study drugs up to 28 days after the last dose of study drugs. Maximum duration between first and last dose: 505 days for Arm A, 414 days for Arm B, 842 days for Arm C, 728 days for Arm B Expansion.
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Participants
  Grade 1 AEs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 AEs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 5 | 0 | 3 | 3 | 1 | 1 | 3
  Grade 3 AEs | 2 | 2 | 2 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 9 | 2 | 2 | 6 | 4 | 4 | 0 | 2 | 8 | 7
  Grade 4 AEs | 2 | 2 | 1 | 2 | 5 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Grade 5 AEs | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Treatment Related) - Arms A, B, C and B Expansion
Description: as for outcome 3
Time Frame: as for outcome 3
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Participants
  Grade 1 AEs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 AEs | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 6 | 1 | 4 | 3 | 1 | 4 | 4
  Grade 3 AEs | 2 | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 9 | 3 | 2 | 4 | 2 | 3 | 0 | 2 | 6 | 6
  Grade 4 AEs | 2 | 2 | 1 | 2 | 5 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Grade 5 AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities by Severity (All Cycles) - Hematology
Description: Laboratory abnormalities were graded per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Following parameters were analyzed for laboratory examination: anemia,hemoglobin increased, platelets, white blood cells, absolute neutrophils,lymphocyte count increased, lymphopenia.
Time Frame: as for outcome 3
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Participants
  Anemia: Grade 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 2 | 2 | 0 | 0 | 0
  Anemia: Grade 1 | 2 | 2 | 1 | 0 | 3 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 6 | 2 | 5 | 0 | 1 | 1 | 0
  Anemia: Grade 2 | 2 | 1 | 2 | 3 | 2 | 3 | 2 | 1 | 2 | 2 | 6 | 2 | 1 | 5 | 1 | 0 | 1 | 2 | 6 | 8
  Anemia: Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
  Anemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 0 | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 9 | 12
  Hemoglobin increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hemoglobin increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 0 | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 9 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
  Lymphocyte count increased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphopenia: Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2
  Lymphopenia: Grade 1 | 1 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 7 | 2 | 2 | 2 | 0 | 3 | 3
  Lymphopenia: Grade 2 | 2 | 1 | 1 | 1 | 4 | 2 | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 6 | 2 | 4 | 1 | 1 | 3 | 4
  Lymphopenia: Grade 3 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 3
  Lymphopenia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute neutrophils: Grade 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 1 | 2 | 3 | 1 | 14 | 4 | 7 | 2 | 3 | 3 | 5
  Absolute neutrophils: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Absolute neutrophils: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3
  Absolute neutrophils: Grade 3 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
  Absolute neutrophils: Grade 4 | 2 | 3 | 1 | 2 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 0 | 1 | 5 | 2 | 3 | 5 | 2 | 1 | 1 | 2 | 0 | 6 | 3 | 1 | 15 | 4 | 6 | 3 | 3 | 7 | 7
  Platelets: Grade 1 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 3
  Platelets: Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White blood cells: Grade 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 2 | 2 | 1 | 10 | 3 | 6 | 1 | 3 | 1 | 1
  White blood cells: Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 3 | 1 | 5 | 1 | 1 | 2 | 0 | 3 | 5
  White blood cells: Grade 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
  White blood cells: Grade 3 | 2 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  White blood cells: Grade 4 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities by Severity (All Cycles) - Coagulation
Description: Laboratory abnormalities were graded per NCI CTCAE version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Following parameters were analyzed for laboratory examination: partial thromboplastin time and prothrombin time international normalized ratio(INR).
Time Frame: as for outcome 3
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Participants
  Partial thromboplastin time: Grade 0 | 4 | 4 | 3 | 2 | 5 | 2 | 3 | 3 | 2 | 2 | 9 | 5 | 2 | 7 | 2 | 4 | 1 | 2 | 9 | 10
  Partial thromboplastin time: Grade 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 6 | 1 | 2 | 1 | 1 | 1 | 1
  Partial thromboplastin time: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
  Partial thromboplastin time: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Partial thromboplastin time: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin time INR: Grade 0 | 1 | 4 | 2 | 3 | 4 | 3 | 3 | 3 | 2 | 3 | 9 | 5 | 2 | 13 | 4 | 6 | 3 | 3 | 8 | 10
  Prothrombin time INR: Grade 1 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
  Prothrombin time INR: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Prothrombin time INR: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin time INR: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities by Severity (All Cycles) - Chemistry
Description: Laboratory abnormalities were graded per NCI CTCAE version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Following parameters were analyzed for laboratory examination: alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), total bilirubin, creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, and hypophosphatemia.
Time Frame: as for outcome 3
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Participants
  ALT: Grade 0 | 3 | 4 | 2 | 2 | 5 | 3 | 2 | 2 | 1 | 2 | 5 | 1 | 0 | 10 | 3 | 6 | 3 | 3 | 7 | 7
  ALT: Grade 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 4 | 2 | 5 | 1 | 1 | 0 | 0 | 2 | 5
  ALT: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALT: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase: Grade 0 | 3 | 4 | 2 | 2 | 4 | 2 | 2 | 1 | 1 | 1 | 8 | 3 | 1 | 9 | 2 | 7 | 3 | 1 | 10 | 8
  Alkaline phosphatase: Grade 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 5 | 1 | 0 | 0 | 2 | 0 | 3
  Alkaline phosphatase: Grade 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Alkaline phosphatase: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Grade 0 | 3 | 2 | 2 | 2 | 4 | 3 | 1 | 2 | 1 | 1 | 9 | 3 | 1 | 12 | 3 | 5 | 3 | 2 | 5 | 6
  AST: Grade 1 | 1 | 3 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 2 | 0 | 1 | 5 | 5
  AST: Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AST: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST: Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 0 | 3 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 9 | 5 | 2 | 13 | 4 | 5 | 3 | 3 | 10 | 12
  Bilirubin (total): Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total): Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Creatinine: Grade 1 | 4 | 5 | 2 | 1 | 4 | 2 | 2 | 3 | 1 | 3 | 6 | 3 | 1 | 12 | 3 | 7 | 3 | 3 | 6 | 4
  Creatinine: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 4 | 5
  Creatinine: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 0 | 4 | 4 | 2 | 2 | 5 | 4 | 3 | 3 | 2 | 3 | 8 | 5 | 2 | 13 | 3 | 7 | 3 | 3 | 8 | 10
  Hypercalcemia: Grade 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 2
  Hypercalcemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia: Grade 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 6 | 1 | 4 | 1 | 2 | 4 | 2
  Hyperglycemia: Grade 1 | 2 | 4 | 1 | 1 | 3 | 3 | 2 | 1 | 0 | 1 | 5 | 3 | 2 | 8 | 2 | 3 | 2 | 0 | 4 | 7
  Hyperglycemia: Grade 2 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Hyperglycemia: Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperglycemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 0 | 4 | 4 | 2 | 1 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 13 | 4 | 7 | 3 | 2 | 9 | 11
  Hyperkalemia: Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
  Hyperkalemia: Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hyperkalemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 0 | 4 | 5 | 2 | 2 | 4 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 6 | 3 | 3 | 10 | 11
  Hypermagnesemia: Grade 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Hypermagnesemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 0 | 4 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
  Hypernatremia: Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 0 | 1 | 4 | 2 | 1 | 3 | 3 | 2 | 3 | 1 | 1 | 6 | 2 | 0 | 9 | 2 | 6 | 2 | 2 | 5 | 10
  Hypoalbuminemia: Grade 1 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 2 | 4 | 2 | 1 | 1 | 1 | 5 | 0
  Hypoalbuminemia: Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Hypoalbuminemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 0 | 1 | 4 | 2 | 2 | 4 | 4 | 0 | 3 | 2 | 2 | 8 | 3 | 1 | 10 | 3 | 6 | 2 | 2 | 9 | 5
  Hypocalcemia: Grade 1 | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 5 | 1 | 1 | 1 | 1 | 0 | 6
  Hypocalcemia: Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Hypocalcemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 0 | 4 | 5 | 3 | 3 | 5 | 3 | 3 | 3 | 2 | 3 | 9 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
  Hypoglycemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 0 | 3 | 5 | 2 | 2 | 5 | 4 | 1 | 2 | 2 | 2 | 3 | 4 | 1 | 11 | 2 | 6 | 2 | 3 | 10 | 7
  Hypokalemia: Grade 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 5 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 2
  Hypokalemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 3
  Hypokalemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia: Grade 0 | 2 | 5 | 3 | 3 | 5 | 2 | 1 | 0 | 1 | 3 | 4 | 2 | 1 | 6 | 0 | 5 | 2 | 2 | 5 | 4
  Hypomagnesemia: Grade 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 3 | 2 | 1 | 9 | 4 | 2 | 1 | 1 | 4 | 5
  Hypomagnesemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Hypomagnesemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hypomagnesemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 0 | 1 | 3 | 2 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 5 | 1 | 0 | 6 | 3 | 4 | 2 | 1 | 6 | 5
  Hyponatremia: Grade 1 | 3 | 1 | 0 | 2 | 3 | 3 | 1 | 2 | 1 | 2 | 4 | 2 | 2 | 6 | 1 | 2 | 1 | 2 | 4 | 6
  Hyponatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1
  Hyponatremia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia: Grade 0 | 1 | 4 | 1 | 0 | 4 | 3 | 1 | 1 | 1 | 2 | 9 | 4 | 1 | 14 | 2 | 5 | 3 | 2 | 8 | 8
  Hypophosphatemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Hypophosphatemia: Grade 2 | 3 | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4
  Hypophosphatemia: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  Hypophosphatemia: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities by Severity (All Cycles) - Urinalysis
Description: Laboratory abnormalities were graded per NCI CTCAE version 4.03 (Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Following parameter was analyzed for laboratory examination: urine protein.
Time Frame: as for outcome 3
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 2 | 10 | 12
Participants
  Grade 0 | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 2 | 0 | 1 | 8 | 5 | 0 | 6 | 4 | 3 | 3 | 1 | 8 | 5
  Grade 1 | 3 | 3 | 2 | 2 | 2 | 1 | 2 | 1 | 3 | 1 | 2 | 0 | 2 | 6 | 0 | 2 | 0 | 0 | 2 | 7
  Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-defined Criteria
Description: Blood pressure (BP), including systolic BP (SBP) and diastolic BP (DBP), and pulse rate were recorded in sitting position.
Time Frame: From baseline up to follow up (at least 28 days and no more than 35 days after discontinuation of treatment). Maximum duration between first and last dose: 842 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3 | 10 | 12
Participants
  Sitting SBP<=100 mmHg | 1 | 2 | 0 | 3 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 2 | 1 | 4 | 1 | 2 | 2 | 0 | 6 | 6
  Sitting SBP>=160 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2
  Sitting DBP<=60 mmHg | 1 | 2 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 2 | 2 | 0 | 5 | 2 | 2 | 1 | 0 | 7 | 6
  Sitting DBP>=100 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting heart rate<50 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting heart rate>120 bpm | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Max increase from baseline in sitting SBP>=20 mmHg | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 4 | 1 | 2 | 3 | 1 | 4 | 1 | 0 | 4 | 4
  Max increase from baseline in sitting SBP>=40 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1
  Max increase from baseline in sitting SBP>=60 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Max increase from baseline in sitting DBP>=10 mmHg | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 2 | 1 | 2 | 8 | 2 | 1 | 4 | 1 | 3 | 1 | 0 | 6 | 5
  Max increase from baseline in sitting DBP>=20 mmHg | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 3
  Max increase from baseline in sitting DBP>=30 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single IV Infusion Dose of PF-05212384 Alone - Plasma PF-05212384 (Arms A, B and C)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose 7 days prior to Cycle 1 Day 1 for Arms A and B; pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose 14 days prior to Cycle 1 Day 1 for Arm C.
Population: All enrolled participants who started treatment and who had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3
ng/mL | 6455 (30) | 9539 (24) | 12090 (21) | 7128 (154) | 12420 (27) | 4522 (76) | 7297 (6) | 7969 (39) | 9548 (20) | 13350 (54) | 15170 (63) | 11510 (61) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 6703 (57) | 8999 (49) | 6783 (24) | 4266 (80) | 8261 (12)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single IV Infusion Dose of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B Expansion)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 (predose Day 8) hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 12
ng/mL | 11340 (60) | 10690 (44)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Docetaxel- Plasma PF-05212384 (Arm A)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 4
ng/mL | 8032 (36) | 8095 (33) | 10380 (26) | 11110 (53) | 10860 (33)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 10 | 4 | 2
ng/mL | 10670 (114) | 7830 (104) | 6273 (102) | 9619 (57) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 18730 (24) | 15000 (19) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Dacomitinib - Plasma PF-05212384 (Arm C)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 13 | 1 | 6 | 3 | 2
ng/mL | 6739 (50) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 6328 (31) | 8547 (48) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B Expansion)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 (predose Day 8) hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 11
ng/mL | 9027 (52) | 14670 (32)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single IV Infusion Dose of Docetaxel Alone- Plasma Docetaxel (Arm A)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5
ng/mL | 946.7 (116) | 2451 (23) | 2528 (19) | 1529 (93) | 1058 (161)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration of Docetaxel IV Infusion in Combination With PF-05212384 - Plasma Docetaxel (Arm A)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 4
ng/mL | 1840 (95) | 695.9 (253) | 2457 (18) | 1424 (126) | 1300 (238)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Single IV Infusion Dose of Cisplatin Alone - Plasma Platinum (Arm B)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 2, 2.5, 3, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2
ng/mL | 3397 (29) | 3950 (1) | 3014 (10) | 4041 (14) | 3337 (8) | 3474 (31) | 3293 (18) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration of Cisplatin IV Infusion in Combination With PF-05212384 - Plasma Platinum (Arm B)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 2, 2.5, 3, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 4 | 2
ng/mL | 3867 (16) | 4201 (7) | 3205 (17) | 4086 (10) | 3130 (17) | 3665 (23) | 3211 (19) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

20. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Multiple Oral Doses of Dacomitinib Alone - Plasma Dacomitinib (Arm C)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 14 | 3 | 7 | 3
ng/mL | 41.04 (33) | 76.24 (45) | 34.17 (61) | 49.90 (38)

21. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Multiple Oral Doses of Dacomitinib in Combination With PF-05212384 - Plasma Dacomitinib (Arm C)
Description: Cmax is defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 12 | 2 | 7 | 3
ng/mL | 52.38 (36) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 33.64 (94) | 48.10 (72)

22. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) Following Single IV Infusion Dose of PF-05212384 Alone - Plasma PF-05212384 (Arms A, B and C)
Description: AUClast is defined as area under the curve from time zero to last quantifiable concentration.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 2 | 4 | 3 | 2 | 4 | 3 | 3 | 1 | 3 | 3 | 8 | 4 | 2 | 14 | 4 | 7 | 3 | 3
ng*hr/mL | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 12530 (26) | 15270 (21) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 18710 (28) | 6756 (65) | 8937 (21) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 14370 (16) | 17710 (14) | 24540 (35) | 24480 (30) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 9191 (32) | 13360 (35) | 10050 (26) | 9493 (32) | 10370 (23)

23. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Docetaxel- Plasma PF-05212384 (Arm A)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: All enrolled participants who started treatment and who have sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 4
ng*hr/mL | 10420 (44) | 15110 (22) | 15520 (26) | 14540 (56) | 15890 (27)

24. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose 7 days prior to Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 1 | 10 | 3 | 2
ng*hr/mL | 14620 (75) | 12690 (58) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 18920 (77) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 38850 (71) | 27480 (46) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 54700 and 69500 ng*hr/mL, respectively.

25. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Dacomitinib - Plasma PF-05212384 (Arm C)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 13 | 1 | 6 | 3 | 2
ng*hr/mL | 10870 (36) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 9977 (22) | 15910 (45) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

26. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Single IV Infusion Dose of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B Expansion)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 (predose Day 8) hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 9 | 12
ng*hr/mL | 20180 (42) | 24480 (22)

27. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B Expansion)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 (predose Day 8) hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 7 | 9
ng*hr/mL | 25250 (49) | 31160 (27)

28. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) Following Single IV Infusion Dose of Docetaxel Alone- Plasma Docetaxel (Arm A)
Description: AUClast is defined as area under the curve from time zero to last quantifiable concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 3 | 5 | 3 | 3 | 5
ng*hr/mL | 1418 (88) | 2748 (27) | 2111 (11) | 1594 (64) | 1280 (63)

29. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) Following Administration of Docetaxel in Combination With PF-05212384 - Plasma Docetaxel (Arm A)
Description: AUClast is defined as area under the curve from time zero to last quantifiable concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 3 | 2 | 3 | 4
ng*hr/mL | 2921 (60) | 2175 (26) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 1415 (115) | 1383 (136)

30. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) Following Single IV Infusion Dose of Cisplatin Alone - Plasma Platinum (Arm B)
Description: AUClast is defined as area under the curve from time zero to last quantifiable concentration.
Time Frame: Pre-dose, 2, 2.5, 3, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2
ng*hr/mL | 50210 (7) | 50860 (6) | 44240 (8) | 48870 (18) | 42910 (23) | 46560 (13) | 48350 (24) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

31. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) Following Administration of Cisplatin IV Infusion in Combination With PF-05212384 - Plasma Platinum (Arm B)
Description: AUClast is defined as area under the curve from time zero to last quantifiable concentration.
Time Frame: Pre-dose, 2, 2.5, 3, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 9 | 4 | 2
ng*hr/mL | 59390 (7) | 62990 (11) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 56170 (22) | 52940 (10) | 53470 (11) | 47500 (18) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

32. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Multiple Oral Doses of Dacomitinib Alone - Plasma Dacomitinib (Arm C)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 13 | 3 | 7 | 3
ng*hr/mL | 818.8 (34) | 1604 (36) | 697.0 (62) | 1040 (34)

33. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to Time Tau (AUCtau) Following Multiple Oral Doses of Dacomitinib in Combination With PF-05212384 - Plasma Dacomitinib (Arm C)
Description: AUCtau is defined as area under the concentration-time profile from time 0 to time tau.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 12 | 2 | 7 | 2
ng*hr/mL | 1069 (38) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 703.8 (100) | NA (NA) — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

34. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Single IV Infusion Dose of PF-05212384 Alone - Plasma PF-05212384 (Arms A, B and C)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2 | 15 | 4 | 7 | 3 | 3
hr | 0.500 [0.500 to 0.567] | 0.500 [0.500 to 0.533] | 0.500 [0.500 to 0.500] | 0.550 [0.517 to 0.833] | 0.500 [0.500 to 0.533] | 0.584 [0.500 to 1.10] | 0.517 [0.500 to 0.533] | 0.500 [0.500 to 0.567] | 0.500 [0.500 to 0.517] | 0.533 [0.500 to 0.617] | 0.509 [0.500 to 1.32] | 0.500 [0.500 to 1.00] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 0.567] | 0.533 [0.500 to 0.700] | 0.500 [0.500 to 0.983] | 0.533 [0.500 to 0.550]

35. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Docetaxel- Plasma PF-05212384 (Arm A)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 4
hr | 0.517 [0.467 to 0.550] | 0.500 [0.500 to 0.833] | 0.500 [0.500 to 0.533] | 0.517 [0.517 to 0.800] | 0.542 [0.500 to 0.583]

36. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 10 | 4 | 2
hr | 0.500 [0.500 to 0.583] | 0.500 [0.500 to 0.533] | 0.550 [0.500 to 1.00] | 0.500 [0.500 to 0.517] | 0.675 [0.600 to 0.750] | 0.517 [0.500 to 2.00] | 0.517 [0.500 to 0.550] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

37. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Dacomitinib - Plasma PF-05212384 (Arm C)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 13 | 1 | 6 | 3 | 2
hr | 0.500 [0.500 to 0.900] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 0.500 [0.500 to 0.600] | 0.500 [0.500 to 0.583] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

38. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Single IV Infusion Dose of Docetaxel Alone- Plasma Docetaxel (Arm A)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5
hr | 1.12 [1.00 to 1.17] | 1.00 [1.00 to 1.50] | 1.00 [1.00 to 1.03] | 1.02 [1.00 to 1.17] | 1.05 [1.00 to 2.05]

39. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Administration of Docetaxel IV Infusion in Combination With PF-05212384 - Plasma Docetaxel (Arm A)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 4
hr | 1.06 [1.00 to 1.13] | 1.34 [1.00 to 2.17] | 1.03 [1.00 to 1.07] | 1.02 [1.02 to 1.02] | 1.13 [1.00 to 1.50]

40. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Single IV Infusion Dose of Cisplatin Alone - Plasma Platinum (Arm B)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 2, 2.5, 3, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2
hr | 2.08 [2.00 to 3.13] | 2.12 [2.02 to 2.23] | 2.10 [2.00 to 2.17] | 2.00 [2.00 to 2.02] | 2.05 [2.00 to 2.08] | 2.01 [1.98 to 2.28] | 2.00 [2.00 to 2.77] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

41. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Administration of Cisplatin IV Infusion in Combination With PF-05212384 - Plasma Platinum (Arm B)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 2, 2.5, 3, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 4 | 2
hr | 2.05 [2.00 to 2.25] | 2.00 [2.00 to 2.03] | 2.00 [2.00 to 2.17] | 2.00 [2.00 to 2.02] | 2.00 [1.62 to 2.50] | 2.02 [1.87 to 2.25] | 2.01 [2.00 to 2.02] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values.

42. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Multiple Oral Doses of Dacomitinib Alone - Plasma Dacomitinib (Arm C)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 14 | 3 | 7 | 3
hr | 4.08 [0.000 to 24.0] | 6.00 [5.92 to 23.3] | 6.00 [4.00 to 25.4] | 5.97 [5.42 to 6.00]

43. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Multiple Oral Doses of Dacomitinib in Combination With PF-05212384 - Plasma Dacomitinib (Arm C)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 12 | 2 | 7 | 3
hr | 6.04 [4.00 to 25.1] | NA [NA to NA] — Summary statistics are not presented if fewer than 3 participants had reportable parameter values. | 6.00 [5.63 to 24.2] | 5.42 [4.00 to 5.50]

44. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Single IV Infusion Dose of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B Expansion)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 (predose Day 8) hours post-dose on Cycle 1 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 12
hr | 0.517 [0.517 to 1.75] | 0.600 [0.500 to 1.25]

45. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Multiple IV Infusion Doses of PF-05212384 in Combination With Cisplatin - Plasma PF-05212384 (Arm B Expansion)
Description: Tmax is defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24, 72, 96 and 168 (predose Day 8) hours post-dose on Cycle 2 Day 1.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 11
hr | 0.517 [0.500 to 1.50] | 0.500 [0.467 to 1.00]

46. Secondary Outcome: Mean Serum Biomarkers for Glucose - Baseline
Description: A phosphatidylinositol 3 kinase/mammalian target of rapamycin (PI3K/mTOR) inhibitor should disrupt the cellular uptake and metabolism of glucose. This study employed metabolic biomarkers such as glucose as pharmacodynamics markers for dual PI3K/mTOR inhibition.
Time Frame: Baseline
Population: The serum pharmacodynamic analysis set was defined as all enrolled participants who started treatment and had a baseline and at least one post baseline measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Arm A: Participants with castrate resistant prostate cancer (CRPC), advanced breast cancer (ABC), or non-small cell lung cancer (NSCLC) that were candidates to treatment with a docetaxel-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90-180 mg once on Day -7 and Cycle 1 Day 2, and docetaxel 75 mg/m2 1-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received docetaxel 75 mg/m2 1-hour IV infusion once followed by PF-05212384 90-180 mg once. The maximum duration of PF-05212384 treatment was 505 days and the maximum duration of docetaxel treatment was 445 days.
- Arm B: Participants with urothelial transitional cell cancer (TCC), triple negative breast cancer (TNBC), NSCLC or ovarian cancer (OC) that were candidates to treatment with a cisplatin-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90-310 mg once on Day -7 and Cycle 1 Day 2, and cisplatin 75 mg/m2 2-hour IV infusion once on Cycle 1 Day 1. On Day 1 for Cycles 2 and beyond, participants received cisplatin 75 mg/m2 2-hour IV infusion once followed by PF-05212384 90-310 mg once. The maximum duration of PF-05212384 treatment was 414 days and the maximum duration of cisplatin treatment was 157 days.
- Arm C: Participants with Her2+ breast cancer (BC) refractory to prior herceptin or lapatinib, Her2+ esophago gastric cancer, head and neck squamous cell cancer (HNSCC), or NSCLC that were candidates to treatment with a dacomitinib-based combination. Each treatment cycle was defined as 21 days. Participants received intravenous infusion of PF-05212384 90-150 mg once on Day -14 and dacomitinib 30-45 mg orally once on Day -7. On Cycle 1 Day 1, participants received dacomitinib 30-45 mg orally once. On Cycle 1 Day 2, participants received treatment with dacomitinib 30 mg orally once followed by PF-05212384 90-150 mg once. On Day 1 for Cycles 2 and beyond, participants received dacomitinib 30-45 mg orally once followed by PF-05212384 90-150 mg once. The maximum duration of PF-05212384 treatment was 842 days and the maximum duration of dacomitinib treatment was 841 days.
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 19 | 32 | 31
mg/dL
  In population of BC: number analyzed (Participants) | 5 | 0 | 5
  In population of BC | 106.80 (18.820) |  | 95.07 (12.019)
  In population of NSCLC: number analyzed (Participants) | 9 | 5 | 8
  In population of NSCLC | 99.56 (15.316) | 100.97 (9.154) | 97.00 (10.10)
  In population of prostate cancer: number analyzed (Participants) | 5 | 0 | 0
  In population of prostate cancer | 124.51 (20.624) |  |
  In population of OC: number analyzed (Participants) | 0 | 2 | 0
  In population of OC |  | 102.71 (15.29) |
  In population of TCC: number analyzed (Participants) | 0 | 7 | 0
  In population of TCC |  | 109.70 (18.335) |
  In population of TNBC: number analyzed (Participants) | 0 | 18 | 0
  In population of TNBC |  | 95.66 (10.659) |
  In population of head and neck cancer: number analyzed (Participants) | 0 | 0 | 12
  In population of head and neck cancer |  |  | 90.68 (14.422)
  In population of oesophageal carcinoma: number analyzed (Participants) | 0 | 0 | 6
  In population of oesophageal carcinoma |  |  | 103.54 (14.970)

47. Secondary Outcome: Mean Serum Biomarkers for Glucose - End of Treatment
Description: A phosphatidylinositol 3 kinase/mammalian target of rapamycin (PI3K/mTOR) inhibitor should disrupt the cellular uptake and metabolism of glucose. This studies employed metabolic biomarkers such as glucose as pharmacodynamics markers for dual PI3K/mTOR inhibition.
Time Frame: End of treatment. Maximum duration between first and last dose: 505 days for Arm A, 414 days for Arm B, 842 days for Arm C, 728 days for Arm B Expansion.
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 15 | 29 | 29
mg/dL
  In population of BC: number analyzed (Participants) | 3 | 0 | 4
  In population of BC | 120.00 (37.242) |  | 99.84 (12.820)
  In population of NSCLC: number analyzed (Participants) | 7 | 4 | 8
  In population of NSCLC | 96.13 (10.500) | 108.11 (10.698) | 97.50 (17.046)
  In population of prostate cancer: number analyzed (Participants) | 5 | 0 | 0
  In population of prostate cancer | 136.91 (59.555) |  |
  In population of OC: number analyzed (Participants) | 0 | 2 | 0
  In population of OC |  | 143.26 (34.404) |
  In population of TCC: number analyzed (Participants) | 0 | 6 | 0
  In population of TCC |  | 100.71 (24.112) |
  In population of TNBC: number analyzed (Participants) | 0 | 17 | 0
  In population of TNBC |  | 108.29 (36.210) |
  In population of head and neck cancer: number analyzed (Participants) | 0 | 0 | 11
  In population of head and neck cancer |  |  | 90.19 (15.367)
  In population of oesophageal carcinoma: number analyzed (Participants) | 0 | 0 | 6
  In population of oesophageal carcinoma |  |  | 1.14 (0.210)

48. Secondary Outcome: Mean Serum Biomarkers for Insulin - Baseline
Description: A phosphatidylinositol 3 kinase/mammalian target of rapamycin (PI3K/mTOR) inhibitor should disrupt the cellular uptake and metabolism of glucose. This studies employed metabolic biomarkers such as insulin as pharmacodynamics markers for dual PI3K/mTOR inhibition.
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: microunits/mL
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 15 | 27 | 23
microunits/mL
  In population of BC: number analyzed (Participants) | 4 | 0 | 5
  In population of BC | 10.93 (3.942) |  | 155.14 (212.916)
  In population of NSCLC: number analyzed (Participants) | 7 | 5 | 4
  In population of NSCLC | 28.61 (56.678) | 710.50 (1346.142) | 11.53 (4.279)
  In population of prostate cancer: number analyzed (Participants) | 4 | 0 | 0
  In population of prostate cancer | 12.65 (13.268) |  |
  In population of OC: number analyzed (Participants) | 0 | 2 | 0
  In population of OC |  | 12.50 (1.980) |
  In population of TCC: number analyzed (Participants) | 0 | 5 | 0
  In population of TCC |  | 20.68 (3.446) |
  In population of TNBC: number analyzed (Participants) | 0 | 15 | 0
  In population of TNBC |  | 81.16 (204.586) |
  In population of head and neck cancer: number analyzed (Participants) | 0 | 0 | 8
  In population of head and neck cancer |  |  | 101.31 (187.285)
  In population of oesophageal carcinoma: number analyzed (Participants) | 0 | 0 | 6
  In population of oesophageal carcinoma |  |  | 338.98 (441.323)

49. Secondary Outcome: Mean Serum Biomarkers for Insulin - End of Treatment
Description: as for outcome 48
Time Frame: as for outcome 47
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: microunits/mL
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 15 | 27 | 23
microunits/mL
  In population of BC: number analyzed (Participants) | 3 | 0 | 4
  In population of BC | 19.17 (8.578) |  | 318.62 (365.374)
  In population of NSCLC: number analyzed (Participants) | 5 | 3 | 3
  In population of NSCLC | 22.34 (20.913) | 832.87 (806.616) | 18.26 (10.559)
  In population of prostate cancer: number analyzed (Participants) | 4 | 0 | 0
  In population of prostate cancer | 13.73 (17.017) |  |
  In population of OC: number analyzed (Participants) | 0 | 2 | 0
  In population of OC |  | 80.30 (81.459) |
  In population of TCC: number analyzed (Participants) | 0 | 4 | 0
  In population of TCC |  | 41.65 (8.505) |
  In population of TNBC: number analyzed (Participants) | 0 | 14 | 0
  In population of TNBC |  | 56.69 (120.565) |
  In population of head and neck cancer: number analyzed (Participants) | 0 | 0 | 7
  In population of head and neck cancer |  |  | 289.32 (606.589)
  In population of oesophageal carcinoma: number analyzed (Participants) | 0 | 0 | 5
  In population of oesophageal carcinoma |  |  | 436.94 (612.108)

50. Secondary Outcome: Mean Serum Biomarkers for Hemoglobin A1c (HbA1c) - Baseline
Description: A phosphatidylinositol 3 kinase/mammalian target of rapamycin (PI3K/mTOR) inhibitor should disrupt the cellular uptake and metabolism of glucose. This studies employed metabolic biomarkers such as hemoglobin A1c (HbA1c) as pharmacodynamics markers for dual PI3K/mTOR inhibition.
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 13 | 26 | 18
Percentage of HbA1c
  In population of BC: number analyzed (Participants) | 3 | 0 | 5
  In population of BC | 7.92 (0.115) |  | 7.00 (1.742)
  In population of NSCLC: number analyzed (Participants) | 6 | 4 | 2
  In population of NSCLC | 7.27 (1.074) | 6.65 (0.931) | 5.13 (0.065)
  In population of prostate cancer: number analyzed (Participants) | 4 | 0 | 0
  In population of prostate cancer | 8.03 (0.465) |  |
  In population of OC: number analyzed (Participants) | 0 | 2 | 0
  In population of OC |  | 7.70 (0.354) |
  In population of TCC: number analyzed (Participants) | 0 | 5 | 0
  In population of TCC |  | 7.65 (0.696) |
  In population of TNBC: number analyzed (Participants) | 0 | 15 | 0
  In population of TNBC |  | 7.18 (1.195) |
  In population of head and neck cancer: number analyzed (Participants) | 0 | 0 | 6
  In population of head and neck cancer |  |  | 7.50 (1.107)
  In population of oesophageal carcinoma: number analyzed (Participants) | 0 | 0 | 5
  In population of oesophageal carcinoma |  |  | 7.00 (1.065)

51. Secondary Outcome: Mean Serum Biomarkers for Hemoglobin A1c (HbA1c) - End of Treatment
Description: as for outcome 50
Time Frame: as for outcome 47
Population: The serum pharmacodynamics analysis set was defined as all enrolled participants who started treatment and had a baseline and at least one post baseline measurement.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 13 | 26 | 18
Percentage of HbA1c
  In population of BC: number analyzed (Participants) | 1 | 0 | 3
  In population of BC | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. |  | 8.39 (1.050)
  In population of NSCLC: number analyzed (Participants) | 5 | 2 | 1
  In population of NSCLC | 7.70 (1.087) | 6.74 (1.572) | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values.
  In population of prostate cancer: number analyzed (Participants) | 3 | 0 | 0
  In population of prostate cancer | 8.42 (1.332) |  |
  In population of OC: number analyzed (Participants) | 0 | 2 | 0
  In population of OC |  | 25.10 (22.698) |
  In population of TCC: number analyzed (Participants) | 0 | 3 | 0
  In population of TCC |  | 7.72 (0.551) |
  In population of TNBC: number analyzed (Participants) | 0 | 14 | 0
  In population of TNBC |  | 7.72 (1.408) |
  In population of head and neck cancer: number analyzed (Participants) | 0 | 0 | 6
  In population of head and neck cancer |  |  | 7.72 (1.012)
  In population of oesophageal carcinoma: number analyzed (Participants) | 0 | 0 | 4
  In population of oesophageal carcinoma |  |  | 7.61 (1.404)

52. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Breast Cancer - Arms A and C
Description: Biopsies were obtained at screening and after drug administration. These samples were analyzed predominantly for phosphoprotein biomarkers indicative of pathway modulation, or for genetic markers correlated to drug sensitivity (eg, emerging KRAS mutation and BRAF mutation). BRAF mutation categories included BRAF mutation status and V600E. KRAS mutation categories included GLY12ALA, GLY12ARG, GLY12ASP, GLY12CYS, GLY12SER, GLY12VAL and GLY13ASP.
Time Frame: Baseline
Population: The molecular profiling tumor analysis set was defined as all enrolled participants who start treatment and had baseline archived tumor biopsy formalin fixed paraffin embedded (FFPE) sample (or fresh FFPE if archived was not available) successfully analyzed for at least one of the selected biomarkers.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A | Arm C
Number analyzed (Participants) | 3 | 5
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0 | 0
  BRAF - BRAF mutaion status (mutation not detected) | 33.3 | 40.0
  BRAF - V600E (mutation detected) | 0 | 0
  BRAF - V600E (mutation not detected) | 66.7 | 40.0
  KRAS - GLY12ALA (mutation detected) | 0 | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0 | 80.0
  KRAS - GLY12ARG (mutation detected) | 0 | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0 | 80.0
  KRAS - GLY12ASP (mutation detected) | 0 | 0
  KRAS - GLY12ASP (mutation not detected) | 100.0 | 80.0
  KRAS - GLY12CYS (mutation detected) | 0 | 0
  KRAS - GLY12CYS (mutation not detected) | 100.0 | 80.0
  KRAS - GLY12SER (mutation detected) | 0 | 0
  KRAS - GLY12SER (mutation not detected) | 100.0 | 80.0
  KRAS - GLY12VAL (mutation detected) | 0 | 0
  KRAS - GLY12VAL (mutation not detected) | 100.0 | 80.0
  KRAS - GLY13ASP (mutation detected) | 0 | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0 | 80.0

53. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Non-Small Cell Lung Cancer - Arms A, B and C
Description: as for outcome 52
Time Frame: Baseline
Population: as for outcome 52
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 7 | 5 | 4
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0 | 0 | 0
  BRAF - BRAF mutaion status (mutation not detected) | 14.3 | 80.0 | 25.0
  BRAF - V600E (mutation detected) | 0 | 0 | 0
  BRAF - V600E (mutation not detected) | 85.7 | 20.0 | 75.0
  KRAS - GLY12ALA (mutation detected) | 0 | 5 | 0
  KRAS - GLY12ALA (mutation not detected) | 85.7 | 100.0 | 100.0
  KRAS - GLY12ARG (mutation detected) | 0 | 0 | 0
  KRAS - GLY12ARG (mutation not detected) | 85.7 | 100.0 | 100.0
  KRAS - GLY12ASP (mutation detected) | 14.3 | 0 | 0
  KRAS - GLY12ASP (mutation not detected) | 71.4 | 100.0 | 100.0
  KRAS - GLY12CYS (mutation detected) | 0 | 0 | 0
  KRAS - GLY12CYS (mutation not detected) | 85.7 | 100.0 | 100.0
  KRAS - GLY12SER (mutation detected) | 0 | 0 | 0
  KRAS - GLY12SER (mutation not detected) | 85.7 | 100.0 | 100.0
  KRAS - GLY12VAL (mutation detected) | 0 | 0 | 0
  KRAS - GLY12VAL (mutation not detected) | 85.7 | 100.0 | 100.0
  KRAS - GLY13ASP (mutation detected) | 0 | 0 | 0
  KRAS - GLY13ASP (mutation not detected) | 85.7 | 100.0 | 100.0

54. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Prostate Cancer - Arm A
Description: as for outcome 52
Time Frame: Baseline
Population: as for outcome 52
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A
Number analyzed (Participants) | 3
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0
  BRAF - BRAF mutaion status (mutation not detected) | 66.7
  BRAF - V600E (mutation detected) | 0
  BRAF - V600E (mutation not detected) | 33.3
  KRAS - GLY12ALA (mutation detected) | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0
  KRAS - GLY12ARG (mutation detected) | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0
  KRAS - GLY12ASP (mutation detected) | 0
  KRAS - GLY12ASP (mutation not detected) | 100.0
  KRAS - GLY12CYS (mutation detected) | 0
  KRAS - GLY12CYS (mutation not detected) | 100.0
  KRAS - GLY12SER (mutation detected) | 0
  KRAS - GLY12SER (mutation not detected) | 100.0
  KRAS - GLY12VAL (mutation detected) | 0
  KRAS - GLY12VAL (mutation not detected) | 100.0
  KRAS - GLY13ASP (mutation detected) | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0

55. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Ovarian Cancer - Arm B
Description: Biopsies were obtained at screening and after drug administration. These samples were analyzed predominantly for phosphoprotein biomarkers indicative of pathway modulation, or for genetic markers correlated to drug sensitivity (eg, emerging KRAS mutation and BRAF mutation). BRAF mutation category was BRAF mutation status. KRAS mutation categories included GLY12ALA, GLY12ARG, GLY12ASP, GLY12CYS, GLY12SER, GLY12VAL and GLY13ASP.
Time Frame: Baseline
Population: as for outcome 52
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm B
Number analyzed (Participants) | 2
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0
  BRAF - BRAF mutaion status (mutation not detected) | 100.0
  KRAS - GLY12ALA (mutation detected) | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0
  KRAS - GLY12ARG (mutation detected) | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0
  KRAS - GLY12ASP (mutation detected) | 0
  KRAS - GLY12ASP (mutation not detected) | 100.0
  KRAS - GLY12CYS (mutation detected) | 50.0
  KRAS - GLY12CYS (mutation not detected) | 50.0
  KRAS - GLY12SER (mutation detected) | 0
  KRAS - GLY12SER (mutation not detected) | 100.0
  KRAS - GLY12VAL (mutation detected) | 0
  KRAS - GLY12VAL (mutation not detected) | 100.0
  KRAS - GLY13ASP (mutation detected) | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0

56. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Transitional Cell Carcinoma - Arm B
Description: as for outcome 52
Time Frame: Baseline
Population: as for outcome 52
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm B
Number analyzed (Participants) | 7
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0
  BRAF - BRAF mutaion status (mutation not detected) | 28.6
  BRAF - V600E (mutation detected) | 0
  BRAF - V600E (mutation not detected) | 71.4
  KRAS - GLY12ALA (mutation detected) | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0
  KRAS - GLY12ARG (mutation detected) | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0
  KRAS - GLY12ASP (mutation detected) | 0
  KRAS - GLY12ASP (mutation not detected) | 100.0
  KRAS - GLY12CYS (mutation detected) | 0
  KRAS - GLY12CYS (mutation not detected) | 100.0
  KRAS - GLY12SER (mutation detected) | 0
  KRAS - GLY12SER (mutation not detected) | 100.0
  KRAS - GLY12VAL (mutation detected) | 14.3
  KRAS - GLY12VAL (mutation not detected) | 85.7
  KRAS - GLY13ASP (mutation detected) | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0

57. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Triple Negative Breast Cancer - Arm B
Description: as for outcome 52
Time Frame: Baseline
Population: The molecular profiling tumor analysis set was defined as all enrolled participants who started treatment and had baseline archived tumor biopsy formalin fixed paraffin embedded (FFPE) sample (or fresh FFPE if archived was not available) successfully analyzed for at least one of the selected biomarkers.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm B
Number analyzed (Participants) | 13
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0
  BRAF - BRAF mutaion status (mutation not detected) | 38.5
  BRAF - V600E (mutation detected) | 0
  BRAF - V600E (mutation not detected) | 38.5
  KRAS - GLY12ALA (mutation detected) | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0
  KRAS - GLY12ARG (mutation detected) | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0
  KRAS - GLY12ASP (mutation detected) | 0
  KRAS - GLY12ASP (mutation not detected) | 100.0
  KRAS - GLY12CYS (mutation detected) | 0
  KRAS - GLY12CYS (mutation not detected) | 100.0
  KRAS - GLY12SER (mutation detected) | 0
  KRAS - GLY12SER (mutation not detected) | 100.0
  KRAS - GLY12VAL (mutation detected) | 0
  KRAS - GLY12VAL (mutation not detected) | 100.0
  KRAS - GLY13ASP (mutation detected) | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0

58. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Head and Neck Cancer - Arm C
Description: as for outcome 52
Time Frame: Baseline
Population: as for outcome 57
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm C
Number analyzed (Participants) | 10
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0
  BRAF - BRAF mutaion status (mutation not detected) | 10.0
  BRAF - V600E (mutation detected) | 0
  BRAF - V600E (mutation not detected) | 90.0
  KRAS - GLY12ALA (mutation detected) | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0
  KRAS - GLY12ARG (mutation detected) | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0
  KRAS - GLY12ASP (mutation detected) | 0
  KRAS - GLY12ASP (mutation not detected) | 100.0
  KRAS - GLY12CYS (mutation detected) | 0
  KRAS - GLY12CYS (mutation not detected) | 100.0
  KRAS - GLY12SER (mutation detected) | 0
  KRAS - GLY12SER (mutation not detected) | 100.0
  KRAS - GLY12VAL (mutation detected) | 0
  KRAS - GLY12VAL (mutation not detected) | 100.0
  KRAS - GLY13ASP (mutation detected) | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0

59. Secondary Outcome: Percentage of Participants With BRAF and KRAS Mutations in Population of Oesophageal Carcinoma - Arm C
Description: as for outcome 52
Time Frame: Baseline
Population: as for outcome 57
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm C
Number analyzed (Participants) | 7
Percentage of Participants
  BRAF - BRAF mutaion status (mutation detected) | 0
  BRAF - BRAF mutaion status (mutation not detected) | 42.9
  BRAF - V600E (mutation detected) | 0
  BRAF - V600E (mutation not detected) | 42.9
  KRAS - GLY12ALA (mutation detected) | 0
  KRAS - GLY12ALA (mutation not detected) | 100.0
  KRAS - GLY12ARG (mutation detected) | 0
  KRAS - GLY12ARG (mutation not detected) | 100.0
  KRAS - GLY12ASP (mutation detected) | 14.3
  KRAS - GLY12ASP (mutation not detected) | 85.7
  KRAS - GLY12CYS (mutation detected) | 0
  KRAS - GLY12CYS (mutation not detected) | 100.0
  KRAS - GLY12SER (mutation detected) | 0
  KRAS - GLY12SER (mutation not detected) | 100.0
  KRAS - GLY12VAL (mutation detected) | 0
  KRAS - GLY12VAL (mutation not detected) | 100.0
  KRAS - GLY13ASP (mutation detected) | 0
  KRAS - GLY13ASP (mutation not detected) | 100.0

60. Secondary Outcome: Number of Participants With Maximum Increase From Baseline in Corrected QT (QTc) Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Participants with maximum increase from baseline of 30 to less than (<) 60 msec(borderline) and greater than or equal to (>=) 60 msec (prolonged) were summarized.
Time Frame: Baseline, Cycle 1 Day 1 (for Arm B Expansion), Cycle 1 Day 2 (for Arms A, B and C), Cycle 2 Day 1 (for Arms A, B and C), Day 1 for each cycle (Cycles 3-36, for Arms B Expansion and C) and end of treatment (up to 2 years, for Arms B Expansion and C).
Population: The QTc analysis set was defined as all enrolled participants who had at least one ECG assessment after receiving study drug or study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 1 | 4 | 4 | 2 | 3 | 1 | 3 | 10 | 4 | 1 | 11 | 2 | 7 | 3 | 2 | 10 | 12
Participants
  Maximum QTcB interval (Bazett's correction) increase from baseline (msec): Change <= 30 | 4 | 5 | 3 | 1 | 4 | 4 | 2 | 3 | 1 | 3 | 10 | 3 | 1 | 10 | 2 | 5 | 3 | 2 | 9 | 7
  Maximum QTcB interval (Bazett's correction) increase from baseline (msec): 30 < Change <= 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4
  Maximum QTcB interval (Bazett's correction) increase from baseline (msec): Change > 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Maximum QTcF interval (Fridericia's correction) increase from baseline (msec): Change <= 30 | 4 | 5 | 3 | 1 | 4 | 4 | 2 | 3 | 1 | 3 | 10 | 3 | 1 | 11 | 2 | 6 | 3 | 2 | 9 | 9
  Maximum QTcF interval (Fridericia's correction) increase from baseline (msec): 30 < Change <= 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Maximum QTcF interval (Fridericia's correction) increase from baseline (msec): Change > 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

61. Secondary Outcome: Number of Participants With Maximum Corrected QT (QTc) Interval Meeting Pre-defined Criteria
Description: QT interval corrected using Fridericia's formula (QTcF) and Bazette's formula (QTcB): QT interval (time corresponding to the beginning of depolarization to re-polarization of the ventricles) divided by cube root of RR interval. Maximum QTcF was categorized as less than (<) 450 milliseconds (msec), 450 msec to 480 msec, 480 msec to 500 msec, and more than (>) 500 msec.
Time Frame: as for outcome 60
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5 | 4 | 3 | 3 | 2 | 3 | 10 | 5 | 2 | 14 | 4 | 7 | 3 | 2 | 10 | 12
Participants
  Maximum QTcB interval (Bazett's correction) (msec): < 450 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 2 | 2 | 2 | 7 | 2 | 2 | 11 | 2 | 5 | 1 | 2 | 5 | 3
  Maximum QTcB interval (Bazett's correction) (msec): 450 <= Value <= 480 | 1 | 2 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 1 | 3 | 3 | 0 | 3 | 2 | 1 | 2 | 0 | 4 | 7
  Maximum QTcB interval (Bazett's correction) (msec): 480 < Value <=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Maximum QTcB interval (Bazett's correction) (msec): > 500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Maximum QTcF interval (Fridericia's correction) (msec): < 450 | 4 | 5 | 3 | 3 | 2 | 4 | 3 | 3 | 2 | 3 | 10 | 4 | 2 | 14 | 4 | 5 | 3 | 2 | 8 | 7
  Maximum QTcF interval (Fridericia's correction) (msec): 450 <= Value <= 480 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
  Maximum QTcF interval (Fridericia's correction) (msec): 480 < Value <=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Maximum QTcF interval (Fridericia's correction) (msec): > 500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

62. Secondary Outcome: Percentage of Participants With Objective Response - Arm A
Description: Percentage of participants with objective response based on the assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm) and no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions.
Time Frame: Baseline up to 18 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 5
Percentage of Participants | 0 [0.0 to 60.2] | 40 [5.3 to 85.3] | 0 [0 to 70.8] | 66.7 [9.4 to 99.2] | 20 [0.5 to 71.6]

63. Secondary Outcome: Percentage of Participants With Objective Response - Arm B
Description: as for outcome 62
Time Frame: Baseline up to 18 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 10 | 5 | 2
Percentage of Participants | 0.0 [0.0 to 60.2] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 20.0 [2.5 to 55.6] | 20.0 [0.5 to 71.6] | 50.0 [1.3 to 98.7]

64. Secondary Outcome: Percentage of Participants With Objective Response - Arm C
Description: as for outcome 62
Time Frame: Baseline up to 18 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm C1: 90 mg PF-05212384 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib
Number analyzed (Participants) | 15 | 4 | 7 | 3 | 3
Percentage of Participants | 20.0 [4.3 to 48.1] | 25.0 [0.6 to 80.6] | 14.3 [0.4 to 57.9] | 0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]

65. Secondary Outcome: Clinical Benefit Response Rate - Arm B Expansion
Description: Percent of participants with confirmed complete response (CR), partial response (PR) or stable disease (SD) for at least 24 weeks on study according to Response Evaluation Criteria in Solid Tumors (RECIST). Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm) and no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions. SD was defined as not qualifying for CR, PR, Progressive Disease (PD).
Time Frame: Baseline up to 18 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 12
Percentage of participants | 60.0 [26.2 to 87.8] | 50.0 [21.1 to 78.9]

66. Secondary Outcome: Duration of Response - Arm B Expansion
Description: Duration of response was calculated from first date of partial response (PR) or complete response (CR) to the date of progression or death due to any cause. In the event of no progression or death, the last tumor assessment date without progression was used in this calculation.
Time Frame: Baseline up to 18 months.
Population: The response analysis set included all participants who received at least one dose of study medication, had the disease under study, had an adequate baseline tumor assessment, and who with objective response.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 4 | 4
month | 6.9 [2.6 to 9.9] | NA [7.4 to NA] — The value marked "NA" was not estimable due to insufficient number of participants with events.

67. Secondary Outcome: Progression Free Survival - Arm B Expansion
Description: Progression free survival (PFS) defined as the time from first dose of study treatment to date of first documentation of progression or death due to any cause, whichever occurs first. PFS was calculated as first event date minus the date of first dose of study medication plus 1 . Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline up to 18 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 10 | 12
month | 4.8 [0.8 to 7.0] | 8.5 [1.2 to NA] — The value marked "NA" was not estimable due to insufficient number of participants with events.

68. Secondary Outcome: Mean Observed Score Values for European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) - Arm B Expansion
Description: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30): included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline, Day 1 and Day 8 of Cycles 1 and 2, Day 1 of Cycles 3 to 16.
Population: All enrolled participants who started treatment on study drug and who completed a baseline assessment and at least one post baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 8 | 11
Score on a scale
  Baseline | 64.58 (18.232) | 58.33 (19.003)
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 10
  Cycle 1 Day 8 | 50.00 (23.570) | 50.00 (26.058)
  Cycle 2 Day 1 | 53.12 (28.499) | 56.82 (17.802)
  Cycle 2 Day 8: number analyzed (Participants) | 7 | 7
  Cycle 2 Day 8 | 50.00 (25.911) | 52.38 (12.468)
  Cycle 3 Day 1: number analyzed (Participants) | 4 | 9
  Cycle 3 Day 1 | 56.25 (38.112) | 57.41 (16.896)
  Cycle 4 Day 1: number analyzed (Participants) | 4 | 9
  Cycle 4 Day 1 | 45.84 (31.551) | 48.15 (19.886)
  Cycle 5 Day 1: number analyzed (Participants) | 5 | 8
  Cycle 5 Day 1 | 45.00 (32.059) | 51.04 (23.753)
  Cycle 6 Day 1: number analyzed (Participants) | 5 | 6
  Cycle 6 Day 1 | 55.00 (33.125) | 51.39 (15.293)
  Cycle 7 Day 1: number analyzed (Participants) | 5 | 6
  Cycle 7 Day 1 | 46.67 (26.745) | 52.78 (20.185)
  Cycle 8 Day 1: number analyzed (Participants) | 5 | 6
  Cycle 8 Day 1 | 51.67 (25.274) | 44.44 (20.860)
  Cycle 9 Day 1: number analyzed (Participants) | 4 | 4
  Cycle 9 Day 1 | 56.25 (20.835) | 56.25 (24.883)
  Cycle 10 Day 1: number analyzed (Participants) | 3 | 4
  Cycle 10 Day 1 | 66.67 (16.665) | 56.25 (15.778)
  Cycle 11 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 11 Day 1 | 54.17 (17.678) | 54.17 (20.971)
  Cycle 12 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 12 Day 1 | 62.50 (29.458) | 52.08 (23.936)
  Cycle 13 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 13 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | 63.89 (17.346)
  Cycle 14 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 14 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | 58.33 (25.000)
  Cycle 15 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 15 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | 61.11 (19.243)
  Cycle 16 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 16 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | 55.56 (9.624)

69. Secondary Outcome: Mean Change From Baseline for European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) - Arm B Expansion
Description: as for outcome 68
Time Frame: Baseline, Day 1 and Day 8 of Cycles 1 and 2, Day 1 of Cycles 3 to 16.
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: 1L Metastasic | Arm 2: 2L/3L Metastatic
Number analyzed (Participants) | 8 | 11
Score on a scale
  Cycle 1 Day 8: number analyzed (Participants) | 4 | 10
  Cycle 1 Day 8 | -16.67 (23.570) | -9.17 (16.411)
  Cycle 2 Day 1 | -11.46 (24.372) | -1.52 (9.734)
  Cycle 2 Day 8: number analyzed (Participants) | 7 | 7
  Cycle 2 Day 8 | -14.28 (26.665) | -7.14 (25.200)
  Cycle 3 Day 1: number analyzed (Participants) | 4 | 9
  Cycle 3 Day 1 | -10.42 (33.591) | 1.85 (18.054)
  Cycle 4 Day 1: number analyzed (Participants) | 4 | 9
  Cycle 4 Day 1 | -14.58 (29.165) | -7.41 (20.601)
  Cycle 5 Day 1: number analyzed (Participants) | 5 | 8
  Cycle 5 Day 1 | -21.67 (34.660) | -5.21 (30.839)
  Cycle 6 Day 1: number analyzed (Participants) | 5 | 6
  Cycle 6 Day 1 | -11.67 (24.719) | -8.33 (22.361)
  Cycle 7 Day 1: number analyzed (Participants) | 5 | 6
  Cycle 7 Day 1 | -20.00 (26.743) | 0.00 (10.545)
  Cycle 8 Day 1: number analyzed (Participants) | 5 | 6
  Cycle 8 Day 1 | -15.00 (18.063) | -8.33 (31.178)
  Cycle 9 Day 1: number analyzed (Participants) | 4 | 4
  Cycle 9 Day 1 | -4.16 (20.971) | -4.16 (22.047)
  Cycle 10 Day 1: number analyzed (Participants) | 3 | 4
  Cycle 10 Day 1 | 5.55 (25.458) | -4.16 (30.808)
  Cycle 11 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 11 Day 1 | 0.01 (23.568) | -6.25 (24.883)
  Cycle 12 Day 1: number analyzed (Participants) | 2 | 4
  Cycle 12 Day 1 | 8.34 (35.348) | -8.34 (32.631)
  Cycle 13 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 13 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | 0.00 (30.044)
  Cycle 14 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 14 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | -5.56 (39.381)
  Cycle 15 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 15 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | -2.78 (29.264)
  Cycle 16 Day 1: number analyzed (Participants) | 1 | 3
  Cycle 16 Day 1 | NA (NA) — Summary statistics are not presented if fewer than 2 participants had reportable parameter values. | -8.33 (22.049)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last treatment administration or until all drug related toxicities have resolved, whichever is later. Maximum duration between first and last dose: 842 days.
Description: Each AE was to be assessed to determine if it met the criteria for SAEs. If an SAE occurred, expedited reporting followed local and international regulations, as appropriate.
Arm/Group | Arm A1: 90 mg PF-05212384 + Docetaxel | Arm A2: 110 mg PF-05212384 + Docetaxel | Arm A3: 130 mg PF-05212384 + Docetaxel | Arm A4: 150 mg PF-05212384 + Docetaxel | Arm A5: 180 mg PF-05212384 + Docetaxel | Arm B1: 90 mg PF-05212384 + Cisplatin | Arm B2: 110 mg PF-05212384 + Cisplatin | Arm B3: 130 mg PF-05212384 + Cisplatin | Arm B4: 150 mg PF-05212384 + Cisplatin | Arm B5: 180 mg PF-05212384 + Cisplatin | Arm B6: 215 mg PF-05212384 + Cisplatin | Arm B7: 260 mg PF-05212384 + Cisplatin | Arm B8: 310 mg PF-05212384 + Cisplatin | Arm C1: 90 mg PF-052123 84 + 30 mg Dacomitinib | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib | Arm 1: 1L Metastatic | Arm 2: 2L/3L Metastatic
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/5 | 0/3 | 1/3 | 0/5 | 0/4 | 0/3 | 1/3 | 0/3 | 1/3 | 0/10 | 1/5 | 0/2 | 0/15 | 2/4 | 0/7 | 0/3 | 0/3 | 0/10 | 1/12
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/5 | 0/3 | 1/3 | 1/5 | 1/4 | 1/3 | 1/3 | 3/3 | 3/3 | 4/10 | 2/5 | 2/2 | 3/15 | 2/4 | 3/7 | 0/3 | 0/3 | 2/10 | 4/12
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 3/3 | 3/3 | 5/5 | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 10/10 | 5/5 | 2/2 | 15/15 | 4/4 | 7/7 | 3/3 | 3/3 | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: 90 mg PF-05212384 + Docetaxel (N=4) | Arm A2: 110 mg PF-05212384 + Docetaxel (N=5) | Arm A3: 130 mg PF-05212384 + Docetaxel (N=3) | Arm A4: 150 mg PF-05212384 + Docetaxel (N=3) | Arm A5: 180 mg PF-05212384 + Docetaxel (N=5) | Arm B1: 90 mg PF-05212384 + Cisplatin (N=4) | Arm B2: 110 mg PF-05212384 + Cisplatin (N=3) | Arm B3: 130 mg PF-05212384 + Cisplatin (N=3) | Arm B4: 150 mg PF-05212384 + Cisplatin (N=3) | Arm B5: 180 mg PF-05212384 + Cisplatin (N=3) | Arm B6: 215 mg PF-05212384 + Cisplatin (N=10) | Arm B7: 260 mg PF-05212384 + Cisplatin (N=5) | Arm B8: 310 mg PF-05212384 + Cisplatin (N=2) | Arm C1: 90 mg PF-052123 84 + 30 mg Dacomitinib (N=15) | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib (N=4) | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib (N=7) | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib (N=3) | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib (N=3) | Arm 1: 1L Metastatic (N=10) | Arm 2: 2L/3L Metastatic (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: 90 mg PF-05212384 + Docetaxel (N=4) | Arm A2: 110 mg PF-05212384 + Docetaxel (N=5) | Arm A3: 130 mg PF-05212384 + Docetaxel (N=3) | Arm A4: 150 mg PF-05212384 + Docetaxel (N=3) | Arm A5: 180 mg PF-05212384 + Docetaxel (N=5) | Arm B1: 90 mg PF-05212384 + Cisplatin (N=4) | Arm B2: 110 mg PF-05212384 + Cisplatin (N=3) | Arm B3: 130 mg PF-05212384 + Cisplatin (N=3) | Arm B4: 150 mg PF-05212384 + Cisplatin (N=3) | Arm B5: 180 mg PF-05212384 + Cisplatin (N=3) | Arm B6: 215 mg PF-05212384 + Cisplatin (N=10) | Arm B7: 260 mg PF-05212384 + Cisplatin (N=5) | Arm B8: 310 mg PF-05212384 + Cisplatin (N=2) | Arm C1: 90 mg PF-052123 84 + 30 mg Dacomitinib (N=15) | Arm C1h: 90 mg PF-05212384 + 45 mg Dacomitinib (N=4) | Arm C2: 110 mg PF-05212384 + 30 mg Dacomitinib (N=7) | Arm C3: 130 mg PF-05212384 + 30 mg Dacomitinib (N=3) | Arm C4: 150 mg PF-05212384 + 30 mg Dacomitinib (N=3) | Arm 1: 1L Metastatic (N=10) | Arm 2: 2L/3L Metastatic (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 2 | 7 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 8 | 11
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 2 | 3 | 5 | 1 | 0 | 0 | 2 | 1 | 5 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 1 | 3 | 0 | 1 | 1 | 1 | 4 | 2 | 2 | 3 | 1 | 2 | 1 | 1 | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 5 | 1 | 1 | 9 | 4 | 6 | 2 | 2 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 1 | 3 | 3 | 2 | 3 | 2 | 2 | 9 | 3 | 2 | 9 | 3 | 4 | 2 | 2 | 7 | 9
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 5
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 8 | 1 | 2 | 6 | 4 | 1 | 1 | 2 | 6 | 8
Asthenia (General disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 5 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 3
Chills (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 1 | 1 | 3 | 2 | 2 | 1 | 3 | 1 | 1 | 5 | 3 | 1 | 9 | 1 | 4 | 1 | 0 | 7 | 9
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 3 | 1 | 2 | 4 | 1 | 1 | 0 | 3 | 1 | 8 | 3 | 2 | 12 | 4 | 6 | 2 | 3 | 6 | 7
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 6 | 5
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 1 | 3 | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 5
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 3 | 0 | 0 | 1 | 4
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 3 | 0 | 1 | 5 | 1 | 0 | 7 | 0 | 2 | 1 | 2 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 4 | 3 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 5 | 4
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 4 | 1 | 1 | 1 | 0 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 8 | 1 | 3 | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 1 | 1 | 3 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 3 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 7 | 2 | 2 | 5 | 0 | 1 | 1 | 0 | 2 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 2 | 4 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ototoxicity (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 6 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cheilosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecthyma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Grip strength decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Human epidermal growth factor receptor decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT01920061/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT01920061/SAP_001.pdf